CLINICAL TRIAL: NCT00945620
Title: Trans-Abdominis Plane Block Efficacy for Post-Cesarean Section Pain: A Randomized Double-Blinded Case Control Trial
Brief Title: Trans-Abdominis Plane Block Efficacy for Post-Cesarean Section Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI was unable to locate appropriate population
Sponsor: Vanderbilt University (Other)
Responsible Party: Sarah A. Starr, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VUMC01TAP; TAP
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Pain Control
Keywords: Trans-abdominis block; post-cesarean
MeSH Terms: conditions — Agnosia | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- right side (Placebo Comparator): The trans-abdominis block will be placed in every pat with one side being injected with ropivicaine, the other side placebo injection. Hence is subject can serve as their own control. Subjects will receive additional pain medications as needed
  Interventions: Drug: placebo
- Left side (Placebo Comparator): The trans-abdominis block will be placed in every pat with one side being injected with ropivicaine, the other side placebo injection. Hence is subject can serve as their own control. Subjects will receive additional pain medications as needed
  Interventions: Drug: ropivicaine

INTERVENTIONS:
Drug: ropivicaine — 30mL containing 300mg ropivicaine 1% with addition of 1:300,000 epinepherine
  Other Names: Trans-Abdominis Plane Block, ropivicaine, naropin
  Arms: Left side
Drug: placebo — Placebo
  Arms: right side

SUMMARY:
The primary aim of this study is to measure the magnitude and duration of trans-abdominis plane (TAP) block analgesia in parturients undergoing elective cesarean section with concurrent standard of care operative analgesic regimens including intrathecal morphine sulfate (ITMS). A one sided block model takes advantage of the bilateral nature of the pain created by a bilateral surgical wound and allows each patient to serve as her own control. Reduced variability allows a more definitive establishment of analgesic benefit for this block.

The current reports of conflicting data regarding efficacy make uncertain the role of TAP block in post cesarean section pain relief. This model would have a better potential for measuring the block's effectiveness. Quantitative sensory evaluation tools such as the von Frey hair tool provides a quantitative reproducible measure of skin sensation and also allows for assessment of block regression over time. Pressure algometry has been established as a clinical and research tool for quantitative assessment of pain levels in multiple pain conditions. A useful inexpensive reliable pressure algometer has recently been described.

The assessment of serum ropivicaine levels with this block will provide useful data regarding the systemic absorption of local anesthetic compared to other peripheral nerve blocks and establish the safety of the technique.

In addition this study will help establish a model for the study of TAP block modifications in the future. If block effectiveness is demonstrated, this model can be used to examine numerous block parameters including choice of local anesthetic and dose response analysis for optimal volume and concentration. Potential future study may be done also in the area of adjuncts found to have increased duration and effectiveness as used in other peripheral nerve blocks.

Expected duration of this study is 18 months.

DETAILED DESCRIPTION:
This will be a randomized, double-blinded prospective trial. Group A patients will be randomized to receive a TAP block with local anesthetic on the right, sham block on the left. Group B be will randomized to receive the reverse. The study population will be limited to healthy parturients undergoing elective caesarian section with spinal anesthesia (SAB) or combined spinal-epidural anesthesia (CSE) placed in the operating room at time of surgery.

Patient recruitment:

Prior to enrollment into the study informed consent will be obtained. Consent will be obtained by a study investigator blinded to the group into which the patient will be randomized. After preanesthetic counseling and patient agreement for a SAB or CSE for cesarean delivery will counsel the patient regarding study participation. Pre-operative instruction of the VAS scale shall be given by the investigator. Routine pre-operative preparations per current protocols will occur.

Intra-operative Anesthetic Regimen:

Anesthetic techniques will be per current protocols. A single intravenous infusion will be used for both intraoperative infusion of intravenous fluids during anesthetic maintenance infusion and for blood sampling for ropivicaine levels following TAP block placement.

SAB and CSE utilizing 12 mg hyperbaric bupivacaine, and 0.15mg intrathecal morphine shall be used as spinal anesthetic for all study patients. Intra-operative conduct of anesthesia will be left to the discretion of anesthesiologist caring for the parturient.

TAP Block Protocol:

At the end of the surgical procedure, if there are no new exclusion criteria, the subject will be randomized to receive bilateral TAP blocks using 30 mL containing 300 mg ropivicaine (1%) with addition of 1:300,000 epinephrine on one side (Group A on the right), and sham needle placement on the other (Group B on the right). During the procedure the study subject shall be blinded to the group assignment by surgical drapes.. The investigator who records the patient assessments will not be present at block placement. The un-blinded anesthesia provider will remove and open 1 of 22 opaque envelopes containing a card identifying the group to which the patient has been assigned by computer generated randomization. The provider will then prepare the injection syringes, labeling the ropivicaine syringe with RIGHT or LEFT according to randomization. The envelope will then be sealed and placed in the patient's study packet. An unblinded investigator trained in the block technique using ultrasound guidance will perform the block.

The TAP block shall be performed in the fashion described by Carney et. al (5). in the region of the triangle of Petit located at the superior aspect of the iliac crest, using a 22g regional block needle, utilizing the 2 pop technique(2) and needle tip position verified by ultrasound imaging. The investigator will confirm placement of the injectate in the fascial plane by initial injection of a small amount of the local anesthetic drug followed by injection of the rest of the dose with ultrasound verification of anesthetic deposition between the internal oblique and transversus abdominis. The ultrasound image will be printed and included with the study data.. The other side will receive a sham needle placement without medication injection. Because this block is performed before regression of spinal anesthesia, it causes no pain to the subject.

Post-Block Care:

Following the placement of the block, all parturients will receive a standard post-operative analgesic regimen that represents our routine practice:

* Toradol 15mg IV upon completion of surgery.
* Percocet 5/325mg q 4 hrs PRN (pain)
* Motrin 600mg q 6 hours PRN (pain)

The time to first analgesic request and administration will be recorded. The total amounts of supplemental analgesics administered will be recorded for the first 48 hours.

Following block placement, venous blood shall be drawn at set intervals described below from the indwelling venous catheter to assess ropivicaine levels.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Pre-pregnancy body mass index less than or equal to 35
* Elective repeat cesarean section under SAB or CSE (patients in whom the epidural catheter is activated intra-operatively will be excluded)
* English-Speaking patient
* Age at least 18 and no more than 40 years old.

Exclusion Criteria:

* Chronic pain or daily consumption of pain medications
* Neurologic disorders producing altered sensory perception or impaired motor strength in lower extremities or abdomen
* Pre-existing epidural analgesia infusion for labor analgesia.
* Spinal anesthetic failure requiring epidural catheter use or general anesthesia
* Intra-operative conversion to general anesthesia for fetal indications.
* Cesarean section performed with a vertical (not Phannenstiel) incision

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Difference in pain perception based upon VAS scores at rest between blocked and unblocked side in each subject | 4, 6, 8, 12, 16, 20 and 24 hours post TAP placement

SECONDARY OUTCOMES:
Difference in pain perception | 4, 6, 8, 12, 16, 20, and 24 hours post TAP
Duration of time at pain perception between sides is equal | 4, 6, 8, 12, 16, 20, and 24 hours post TAP
Duration of time skin sensation of touch | 4, 6, 8, 12, 16, 20, and 24 hours post TAP
Assessment of ropivacaine levels | 4, 6, 8, 12, 16, 20, and 24 hours post TAP

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States